CLINICAL TRIAL: NCT03072446
Title: Uterine Fibroid Embolization (UFE) for Symptomatic Fibroids: Comparison of Gel-Bead to Commonly Used Embolic Agents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Vascular Solutions LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHM RAD0041
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Uterine Fibroid; Embolization; Symptoms
Keywords: Uterine Fibroid; Embolization; symptoms; Gel-Beads
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Gel-Beads arm (Experimental): This group will undergo embolization of symptomatic uterine fibroids with Gel-Beads embolic agent
  Interventions: Device: Gel-Beads embolic material

INTERVENTIONS:
Device: Gel-Beads embolic material — Patients will receive embolization of their uterine fibroids using Gel-Beads.

SUMMARY:
The purpose of this post-market study is to evaluate UFE agents for the treatment of symptomatic uterine fibroids, using Gel-Bead compared to four other commonly used embolic agents.

DETAILED DESCRIPTION:
This single-center, prospective study will be conducted at one site in the United Kingdom. Up to 30 subjects will be enrolled and treated with Gel-Bead. Prospectively. Enrolled Gel-Bead subjects will be followed at 1-month and 3-months post-procedure.

Data from subjects treated with Gel-Bead will be compared to data from a previously unpublished, but widely presented, 100-patient cohort study at the University Hospital Southampton. This study evaluated 20 subjects in five different treatment groups for the treatment of symptomatic uterine fibroids. The five treatment groups include gelatin foam slurry, Embospheres, polyvinyl alcohol (PVA), Bead Block and Embozenes.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age 18 years or older
2. Symptomatic uterine fibroid(s) requiring treatment per the investigators assessment
3. Negative serum pregnancy test at the Baseline visit and practicing effective contraception during the study
4. Willing to provide written informed consent prior to initiation of study procedures
5. Willing to comply with the specified study assessments and follow-up requirements

Exclusion Criteria:

1. Known hypersensitivity to porcine products or intravascular contrast material
2. Vascular anatomy or blood flow precluding correct catheter placement or embolic injection
3. Presence of collateral vessel pathways potentially endangering normal territories during embolization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Degree of Fibroid Tissue Infarction at 3 months | 3 months
  The primary endpoint is the degree of fibroid tissue infarction at 3 months post-procedure. Results for the total fibroid load and the dominant fibroid will be categorized as either 100% (Group A) ≥ 90-99% (Group B) or <90% (Group C) infarcted. The degree of infarction will be visually estimated by the investigator.
Characterization of adverse events over 3 months | 3 months
  The primary safety endpoint is to characterize adverse events

SECONDARY OUTCOMES:
Change in uterine and dominant fibroid volumes | 3 months
  Changes in uterine and dominant fibroid volumes between pre-procedure and Month 3 based on CE-MRI. The absolute dimensions of the uterus will be measured and the approximate uterine volumes will be calculated using the formula for a prolate ellipse (length X width X depth X 0.5233).

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Hacking, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Southampton University Hospital NHS Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers.